CLINICAL TRIAL: NCT05722262
Title: A Randomized, Open-Label, Six-Sequence, Three-Period Crossover Study to Demonstrate the Bioequivalence of Single Oral Administration of K-001 Relative to Single Oral Coadministration of Separate Tablets of K-877-ER Plus CSG452 in Healthy Adult Volunteers, and to Characterize the Food Effect on the Pharmacokinetics of K-001
Brief Title: Study to Demonstrate the Bioequivalence of Single Oral Administration of K-001 Relative to Single Oral Coadministration of Separate Tablets of K-877-ER and CSG452
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: K-001-1.02
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — 6-((4-ethylphenyl)methyl)-3',4',5',6'-tetrahydro-6'-(hydroxymethyl)spiro(isobenzofuran-1(3H),2'-(2H)pyran)-3',4',5'-triol

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, six-sequence, three-period, crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence A (Experimental): Three period alternative intervention and fed/fasted sequence
  Interventions: Drug: K-001; Drug: K-877-ER; Drug: CSG452
- Sequence B (Experimental): Three period alternative intervention and fed/fasted sequence
  Interventions: Drug: K-001; Drug: K-877-ER; Drug: CSG452
- Sequence C (Experimental): Three period alternative intervention and fed/fasted sequence
  Interventions: Drug: K-001; Drug: K-877-ER; Drug: CSG452
- Sequence D (Experimental): Three period alternative intervention and fed/fasted sequence
  Interventions: Drug: K-001; Drug: K-877-ER; Drug: CSG452
- Sequence E (Experimental): Three period alternative intervention and fed/fasted sequence
  Interventions: Drug: K-001; Drug: K-877-ER; Drug: CSG452
- Sequence F (Experimental): Three period alternative intervention and fed/fasted sequence
  Interventions: Drug: K-001; Drug: K-877-ER; Drug: CSG452

INTERVENTIONS:
Drug: K-001 — K-877-ER and CSG452 combination tablet
Drug: K-877-ER — K-877-ER tablet
Drug: CSG452 — CSG452 tablet

SUMMARY:
The goal of this clinical trial is to demonstrate the bioequivalence of single oral administration of K-001 relative to single oral co-administration of separate tablets of K-877-ER and CSG452 in healthy adult volunteers, and to characterize the food effect on the Pharmacokinetics(PK) of K-001.

ELIGIBILITY:
Inclusion Criteria:

* Participant provides written informed consent before any study-specific evaluation is performed.
* Participant is a healthy adult male or female volunteer between the ages of 18 and 45 years, inclusive, at Screening.
* Participant has a body mass index of 18 to 30 kg/m2, inclusive, at Screening.
* Participant meet all other inclusion criteria outlined in the clinical study protocol.

Exclusion Criteria:

* Participant has clinically significant abnormalities at Screening or at Check-in assessments, in the opinion of the investigator.
* Participant is pregnant or breastfeeding or intends to become pregnant within 30 days after the last dose of study drug.
* Participant meets any other exclusion criteria outlined in the clinical study protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Cmax of K-877 and CSG452 | 1 hour before dosing and at multiple time points (up to 48 hours) post dose
  Maximum observed plasma concentration (Cmax) of K-877 and CSG452
AUC0-t of K-877 and CSG452 | 1 hour before dosing and at multiple time points (up to 48 hours) post dose
  Area under the plasma concentration versus time curve from time 0 to the time of the last quantifiable concentration (AUC0-t)
AUC0-inf of K-877-and CSG452 | 1 hour before dosing and at multiple time points (up to 48 hours) post dose
  Area under the plasma concentration versus time curve from time 0 extrapolated to infinity (AUC0-inf).

CONTACTS AND LOCATIONS:
Locations (1):
- PPD - Austin Research Unit, Austin, Texas, United States